CLINICAL TRIAL: NCT02531503
Title: Predicting Factors for Asthma Remission in Children
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, JITTIMA VESKITKUL, Asst.Prof., Mahidol University
Other Study IDs: 697/2557(EC3)
Record Dates: First submitted 2015-08-19; First posted 2015-08-24 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma remission; Predicting factors; Children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical asthma remission: Clinical asthma remission was defined as having no asthma symptoms and no use of asthma medication during the past 12 months.
  Interventions: Other: Clinical asthma remission

INTERVENTIONS:
Other: Clinical asthma remission — Clinical asthma remission was defined as having no asthma symptoms and no use of medication during the past 12 months.

SUMMARY:
The purpose of this study is to determine the predicting factors for asthma remission in children.

DETAILED DESCRIPTION:
Children who were diagnosed as having asthma during the period of 2004-2007 and reevaluated in 2015.

ELIGIBILITY:
Inclusion Criteria:

* Children who were diagnosed as having asthma during the period of 2004-2007.

Exclusion Criteria:

* Patients who had underlying disease with chronic respiratory disease (ex. tuberculosis, bronchiectasis), primary immunodeficiency, other seriously interfering diseases
* Medical records have been lost.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The children who were diagnosed as having asthma at pediatric allergy clinic were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of factors associated with asthma remission | 18 months

SECONDARY OUTCOMES:
Asthma remission rate | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Division of Allergy and Immunology, Department of Pediatrics,, Principal Investigator — Mahidol University
Locations (1):
- Division of Allergy and Immunology, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No